CLINICAL TRIAL: NCT03527485
Title: Imaging Synaptic Density in Cocaine and Opiate Addiction In Vivo Using 11UCB-J PET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2000021843; 1R21DA046030-01A1 (NIH)
Record Dates: First submitted 2018-04-19; First posted 2018-05-17 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-06

CONDITIONS: Opiate Dependence; Cocaine Dependence
MeSH Terms: conditions — Opioid-Related Disorders; Cocaine-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opiate Use Disorder (OUD) (Other): 30 subjects meeting opiate dependence criteria will receive 11UCB-J PET Scan.
  Interventions: Diagnostic Test: 11UCB-J PET Scan
- Healthy Controls (HC) (Other): 30 healthy controls; no substance dependence or mental health issues 11UCB-J PET Scan.
  Interventions: Diagnostic Test: 11UCB-J PET Scan

INTERVENTIONS:
Diagnostic Test: 11UCB-J PET Scan — 11UCB-J PET Scan

SUMMARY:
This study aims to measure synaptic density in the brains (including in ventral striatum [VS] and medial prefrontal cortex [mPFC]) of abstinent subjects with Cocaine Use Disorder (CUD) or Opiate Use Disorder (OUD) as compared to healthy control (HC) subjects using 11C-UCB-J PET. Subjects will undergo a single 11C-UCB-J (also known as 11C-APP311) PET scan.

This would be the very first to image synaptic density in human cocaine and opiate users, thereby testing whether altered synaptic density in the rodent brain is recapitulated in CUD and OUD humans. If confirmed, the current study would provide compelling clinical-translational support for an important pathophysiological mechanism of addiction - aberrant structural synaptic plasticity. As such, the current study has considerable potential for advancing the neurobiological understanding of human cocaine and opiate addiction.

DETAILED DESCRIPTION:
This study aims to measure synaptic density in the brains (including in ventral striatum [VS] and medial prefrontal cortex [mPFC]) of abstinent subjects with Cocaine Use Disorder (CUD) or Opiate Use Disorder (OUD) as compared to healthy control (HC) subjects using 11C-UCB-J PET. Subjects will undergo a single 11C-UCB-J (also known as 11C-APP311) PET scan.

This would be the very first to image synaptic density in human cocaine and opiate users, thereby testing whether altered synaptic density in the rodent brain is recapitulated in CUD and OUD humans. If confirmed, the current study would provide compelling clinical-translational support for an important pathophysiological mechanism of addiction - aberrant structural synaptic plasticity. As such, the current study has considerable potential for advancing the neurobiological understanding of human cocaine and opiate addiction.

A separate protocol from the study team, identified by the ClinicalTrials.gov ID NCT04721418, is conducting a comprehensive investigation into the cocaine use disorder group. Therefore, data for participants with cocaine use disorder are not included in the results for the current registration.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-55 years;
* Voluntary, written, informed consent;
* Physically healthy by medical history, physical, neurological, ECG and laboratory examinations;
* DSM-5 criteria for Opiate Use Disorder;
* Documented evidence (by urine toxicology) of 2 weeks abstinence from cocaine and 4 weeks abstinence from opiates;
* For females, a negative serum pregnancy (HCG) test;
* Full scale and verbal IQs > 80 (Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV)).

Exclusion Criteria:

* A history of other substance dependence (e.g., alcohol, sedative hypnotics), except for nicotine;
* A primary DSM-5 Axis I major psychiatric disorder (e.g., schizophrenia, bipolar disorder, major depression, etc.) as determined by the Structured Clinical Interview for DSM-5 (SCID-5);
* A history of significant and uncontrolled medical (e.g., cardiovascular, diabetic/metabolic) or neurological (e.g., cerebrovascular, seizures, traumatic brain injury) illness;
* A history of seizures;
* Current use of psychotropic and/or potentially psychoactive prescription medications;
* Medical contraindications to participation in a magnetic resonance (MR) imaging procedure (e.g., ferromagnetic implants/foreign bodies, claustrophobia, cardiac pacemaker, prosthetic valve, otologic implant, etc.) as recorded on the MR safety sheet;
* For females, physical or laboratory (HCG) evidence of pregnancy;
* PTT and PT/INR lab results not appropriate for arterial line placement;
* Taking anticoagulants;
* Being prescribed methadone/buprenorphine upon screening.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CT Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Innis RB, Cunningham VJ, Delforge J, Fujita M, Gjedde A, Gunn RN, Holden J, Houle S, Huang SC, Ichise M, Iida H, Ito H, Kimura Y, Koeppe RA, Knudsen GM, Knuuti J, Lammertsma AA, Laruelle M, Logan J, Maguire RP, Mintun MA, Morris ED, Parsey R, Price JC, Slifstein M, Sossi V, Suhara T, Votaw JR, Wong DF, Carson RE. Consensus nomenclature for in vivo imaging of reversibly binding radioligands. J Cereb Blood Flow Metab. 2007 Sep;27(9):1533-9. doi: 10.1038/sj.jcbfm.9600493. Epub 2007 May 9. PMID 17519979

RESULTS

PARTICIPANT FLOW:
Groups:
- Opiate Use Disorder (OUD): 15 subjects meeting opiate dependence criteria will receive 11UCB-J PET Scan.
  11UCB-J PET Scan: 11UCB-J PET Scan
- Healthy Controls (HC): 26 healthy controls; no substance dependence or mental health issues 11UCB-J PET Scan.
  11UCB-J PET Scan: 11UCB-J PET Scan
Period: Overall Study
Arm/Group | Opiate Use Disorder (OUD) | Healthy Controls (HC)
Started | 15 | 26
Completed | 15 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Opiate Use Disorder (OUD) | Healthy Controls (HC) | Total
Number analyzed (Participants) | 15 | 26 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (6.5) | 36.7 (10.6) | 37.0 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 10 | 19 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White (Non-Hispanic) | 15 | 22 | 37
  African American/Black (Non-Hispanic) | 0 | 0 | 0
  Hispanic or Latino | 0 | 2 | 2
  Other or Unknown | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 15 | 26 | 41

OUTCOME MEASURES:

1. Primary Outcome: 11C-UCB-J PET Synaptic Density
Description: PET scan- Participants underwent a single 11C-UCB-J PET scan to obtain measures of synaptic density (BPND). Structural magnetic resonance imaging (MRI) scans were also obtained for anatomical registration/partial volume correction (PVC) with the iterative Yang (IY) algorithm. BPND is a unitless metric. The study aimed to explore synaptic density differences in subjects with opioid use disorder compared to a control group within the sample.
Time Frame: 90 minute scan
Population: All participants who underwent 11C-UCB-J PET and MRI scans
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Opiate Use Disorder (OUD) | Healthy Controls (HC)
Number analyzed (Participants) | 15 | 26
unitless
  Region of Interest: Ventral Striatum (VS) | 4.01 (0.70) | 4.52 (0.53)
  Region of Interest: Prefrontal Cortex (PFC) | 4.62 (0.87) | 5.09 (0.61)
Statistical Analysis 1: Comparison: Opiate Use Disorder (OUD) vs Healthy Controls (HC); Test type: Equivalence — Between-group comparisons of binding potential non displaceable (BPND) in ventral striatum (VS); p = 0.011, ANOVA
Statistical Analysis 2: Comparison: Opiate Use Disorder (OUD) vs Healthy Controls (HC); Test type: Equivalence — Between-group comparisons of binding potential non displaceable (BPND) in Prefrontal cortex (PFC); p = 0.044, ANOVA

ADVERSE EVENTS:
Time Frame: 90 minutes
Arm/Group | Opiate Use Disorder (OUD) | Healthy Controls (HC)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/26
Other Adverse Events (participants affected / at risk) | 0/15 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT03527485/Prot_SAP_000.pdf